CLINICAL TRIAL: NCT06540105
Title: Leveraging Artificial Intelligence and Multi-Omics Data to Predict Opioid Addiction
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rodney Gabriel, Associate Professor, University of California, San Diego
Other Study IDs: 810491
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Opioid Use Disorder; Addiction, Opioid
Keywords: genomics; artificial intelligence; microbiome; opioid use disorder; opioid addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva for DNA sequencing, stool sample for microbiome analyses and blood/plasma for metabolomic analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Opioid Use Disorder: Subjects with a history of opioid use disorder

SUMMARY:
The primary goal of this proposal is to validate a novel genomic and microbiome predictive model that may be used to assess a person's risk of developing opioid use disorder (OUD). The following will be tested: (1) MODUS (Measuring risk for Opioid use Disorder Using SNPs), which is a genomic panel consisting of a set number of proven single nucleotide polymorphisms (SNP) that utilizes machine learning to determine an individual's risk; and (2) MICROUD (MICRObiome for Opioid Use Disorder), which will be a novel microbiome prediction panel for OUD risk. MODUS and MICROUD will be developed using existing public datasets with genomic and microbiome data (e.g., All of Us, Human Microbiome Project). During development of these predictive models, in parallel, an external prospective validation cohort will be recruited consisting of subjects from the University of California, San Diego, Veteran Affairs of San Diego, and Veteran Affairs of Palo Alto (each site with separate IRB). The hypothesis is that MODUS and MICROUD will have high predictive potential for identifying high risk patients for OUD.

DETAILED DESCRIPTION:
The primary goal of this proposal is to validate a novel genomic and microbiome predictive model that may be used to assess a person's risk of developing opioid use disorder (OUD). The following will be tested: (1) MODUS (Measuring risk for Opioid use Disorder Using SNPs), which is a genomic panel consisting of a set number of proven single nucleotide polymorphisms (SNP) that utilizes machine learning to determine an individual's risk; and (2) MICROUD (MICRObiome for Opioid Use Disorder), which will be a novel microbiome prediction panel for OUD risk. MODUS and MICROUD will be developed using existing public datasets with genomic and microbiome data (e.g., All of Us, Human Microbiome Project). During development of these predictive models, in parallel, an external prospective validation cohort will be recruited consisting of subjects from the University of California, San Diego, Veteran Affairs of San Diego, and Veteran Affairs of Palo Alto (each site with separate IRB). The hypothesis is that MODUS and MICROUD will have high predictive potential for identifying high risk patients for OUD.

Specific Aim 1. Validate a novel genomic predictive panel assay - termed MODUS - in a prospective observational study that aims to recruit 300 subjects (~200 from UCSD and VA San Diego) with a history of OUD. This genomic panel will be developed separately but then validated on the study population. Healthy control data will be used from a publicly-available de-identified genomic dataset (All of Us Research Program) .

Specific Aim 2. Validate a novel microbiome predictive panel assay - termed MICROUD - in a prospective observational study that aims to recruit 300 subjects (~200 from UCSD and VA San Diego) with a history of OUD. This microbiome panel will be developed separately but then validated on the study population. Healthy control data will be used from a publicly-available de-identified microbiome dataset (Human Microbiome Project).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OUD (active or in remission) defined by the DSM-5 criteria
* age ≥ 18 years old

Exclusion Criteria:

* inability to participate independently with the study (i.e. dementia)
* chronic opioid use that is not consistent with a diagnosis of OUD
* patients that are pregnant
* children
* institutionalized individuals
* non-English speaking subjects as there are several surveys without appropriate translation and with sensitive information (e.g., questions about mental health and history of drug use) that is required to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the prospective observational study described , adult subjects (≥18 years old) will be recruited with active or previous history of opioid addiction from various clinical settings, including chronic pain clinics, emergency department, operating room, addiction clinics, family medicine/primary care clinics, and surgical clinics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-06-29 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
opioid use disorder at baseline based on the DSM-5 criteria | baseline
  risk of opioid use disorder based on genomics, social determinants of health, microbiome, and other clinical data. Patients with OUD will be enrolled and compared to healthy controls using data from external datasets such as NIH All of Us Research Program. Diagnosis of opioid use disorder will be based on the DSM-5 criteria for opioid use disorder

SECONDARY OUTCOMES:
response to opioid use disorder treatment after 6 months from baseline based on the DSM-5 criteria | 6 months
  prediction of response to opioid use disorder treatment. Remission from opioid use disorder will be based on DSM-5 criteria for remission from substance use disorder
opioid use disorder remission after 6 months from baseline based on the DSM-5 criteria for remission | 6 months
  prediction of remission of opioid use disorder based on the DSM-5 criteria for remission from substance use disorder
severity of opioid use disorder at baseline based on the DSM-5 criteria for opioid use disorder | baseline
  prediction of severity of opioid use disorder based on the DSM-5 criteria for opioid use disorder
co-substance use at baseline | baseline
  risk of developing co-substance use disorder based on DSM-5 criteria for substance use disorders
Relapse to opioid use disorder after 6 months from baseline | 6 months
  risk of relapse to opioid use disorder based on DSM-5 criteria for opioid use disorder

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A Gabriel, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A publicly available biobank with be developed with de-identified data that may be shared with external researchers after approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after conclusion of the study for indeterminate amount of time
Access Criteria: appropriate data use agreement and IRB approval